CLINICAL TRIAL: NCT00474552
Title: An Ascending Multiple-Dose Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of SAM-315 Administered Orally to Healthy Young Adult and Elderly Subjects
Brief Title: Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of SAM-315
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3182A1-101
Record Dates: First submitted 2007-05-15; First posted 2007-05-17 (Estimated); Last update posted 2008-02-18 (Estimated); Status verified 2008-02

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — 3-(naphthalen-1-ylsulfonyl)-5-(piperazin-1-yl)-1H-indazole

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- 1 (Experimental): Experimental-Placebo Comparator
  Interventions: Drug: SAM-315

INTERVENTIONS:
Drug: SAM-315 — Multiple Ascending Doses of SAM-315 (treatment duration: 14 days): 0.2 mg; 0.5 mg; 1 mg; 2 mg;

SUMMARY:
Primary: To assess the safety and tolerability of ascending multiple oral doses of SAM-315, an investigational drug, in healthy young adult and elderly subjects.

Secondary: To assess the Pharmacokinetic and Pharmacodynamic profiles of multiple oral doses of SAM-315 in healthy young adult and elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

Young healthy subjects:

* Men and women of nonchildbearing potential (WONCBP) aged 18 to 45 years inclusive on study day 1.
* Body mass index (BMI) in the range of 18 to 30 kg/m2 and body weight greater than or equal to 50 kg and body weight greater than or equal to 50 kg.

Elderly Healthy subjects:

* Men or women aged 65 years and above as of study day 1.
* BMI in the range of 18 to 30 kg/m2 and body weight greater than or equal to 45 kg and body weight greater than or equal to 45 kg.

Exclusion Criteria:

* Any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease.
* History of any clinically important drug allergy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2007-06; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
safety, tolerability and PK | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For France: infomedfrance@wyeth.com
Locations (1):
- Paris, France